CLINICAL TRIAL: NCT04058041
Title: Effectiveness of Neural Mobilizations Exercises Versus Surgery in Patients With Carpal Tunnel Syndrome
Brief Title: Neural Exercises vs Surgery in Patients With Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPMP/ICH/135/95
Record Dates: First submitted 2018-02-13; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Neuropathic Pain
Keywords: Neural mobilization; Surgery; Pain modulation
MeSH Terms: conditions — Neuralgia | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neural mobilization (Experimental): passive mobilization of the median nerve by the therapist following by an active movement of the fingers of the pathology hand
  Interventions: Procedure: Surgery; Procedure: Surgery and neural mobilization
- Surgery (Active Comparator): the surgeon will release the median nerve in the tunnel carpal. After that the therapist will teach home exercises (no neural exercises) to the patients.
  Interventions: Procedure: Neural Mobilization; Procedure: Surgery and neural mobilization
- Surgery and Neural mobilization (Active Comparator): the surgeon will release the median nerve in the tunnel carpal. After that the therapist will perform mobilizations of the median nerve just like the experimental group.
  Interventions: Procedure: Neural Mobilization; Procedure: Surgery

INTERVENTIONS:
Procedure: Neural Mobilization — neural exercise Will be performed in the patients
  Arms: Surgery; Surgery and Neural mobilization
Procedure: Surgery — open or endoscopic surgery will be permed in the patients with tunnel carpal syndrome
  Arms: Neural mobilization; Surgery and Neural mobilization
Procedure: Surgery and neural mobilization — following the surgery patients will be treat with neural mobilization exercises.
  Arms: Neural mobilization; Surgery

SUMMARY:
neural exercise in patients with carpal tunnel syndrome

DETAILED DESCRIPTION:
OBJECTIVE: The aim objective is to compare the neurophysiological effects of the surgery versus neural mobilization exercises added to surgery versus only neural mobilization exercises on temporal summation and noxious inhibitory pain system and their relationship with the improve of symptoms, with pain and disability in patients with Carpal tunnel syndrome.

STUDY DESIGN: Randomized parallel-group trial. BACKGROUND: Carpal tunnel syndrome (CTS) such as a neuropathic pain condition with altered pain modulation and wind-up, but there is a clack of knowledge if some therapies could have a positive effect.

METHODS: In the Humans study, 54 patients with CTS will be randomly allocated to either a surgery group (n=18) or Surgery with neural exercises group (n=18) or neural exercise group (n=18), the groups with neural exercise will received 10 sessions. The primary outcome will be conditioned pain modulation, temporal summation, pain intensity,. Secondary outcomes will be hand disability assessed with the Boston Carpal Tunnel Questionnaire, pinch-tip grip force, and the symptom severity subscale of the Boston Carpal Tunnel Questionnaire, neuropathic pain questionnaire (DN4), psychological questionnaires (anxiety, catastrophizing, kinesiophobia depression and fear avoid questionnaires), and pressure pain threshold. Patients will be assessed baseline and post-treatment, 1, 3 and 6 months after the last treatment by an assessor unaware of group assignment Patients were assessed at. Analysis was by intention to treat, with mixed analyses of covariance adjusted for baseline scores.

ELIGIBILITY:
Inclusion Criteria:

Tinel and Phalen positive 4/10 in VAS Scale Increase symptoms at night 12 months of symptomatology Sensorial and motor dysfunction in the conduction of the median nerve

Exclusion Criteria:

Previous surgery Wrist fractures Rheumatoid Arthritis or Fibromyalgia Systemic disease Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-02-12 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Physiological parameter | Change from Baseline Conditioned pain modulation at 6 months
  Conditioned pain modulation: Diffuse noxious inhibitory control system will be measure with tourniquet test

SECONDARY OUTCOMES:
Neuropathic pain | Baseline and 6 months
  Neuropathic pain Questionnaire DN4
Pain intensity | Baseline and 6 months
  Visual analog scale. A 100mm VAS, ranging from 0mm (no pain) to 100mm (worst imaginable pain).
Pain expansion | Change from baseline and 6 months
  Body pain maps
Pressure pain threshold | Baseline and 6 months
  Three consecutive trials of pressure pain threshold on the active trigger point at a rate of 1 kg/sec at intervals of 30 seconds were conducted.
Psychological factors_Anxiety | Baseline and 6 months
  State Trait Anxiety Inventory (STAI-T)
Psychological factors_Depression | Baseline and 6 months
  Beck Depression Inventory (BDI-II)
Psychological factors_Kinesiophobia | Baseline and 6 months
  Tampa Scale for Kinesiophobia.. The score goes from 11 to 44. A higher value indicates a worse outcome.
Psychological factors_catastrophizing | Baseline and 6 months
  Pain Catastrophizing Scale. The scores goes from 0 to 52. A higher value indicates a worse outcome.
Psychological factors_Fear avoidance | Baseline and 6 months
  Fear Avoidance Belief Questionnaire (FABQ)
Disability_DASH | Baseline and 6 months
  Disabilities of Arm, Shoulder and Hand (DASH)
Disability_BOSTON | Baseline and 6 months
  Boston Carpal Tunnel Questionnaire
Strength_grip | Baseline and 6 months
  grip strength without pain
Strength_pinch | Baseline and 6 months
  pinch strength

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain